CLINICAL TRIAL: NCT04554732
Title: A Study to Investigate Keratinocyte Growth Factor- Hair Serum for the Prevention of Chemotherapy Induced Alopecia
Brief Title: Keratinocyte Growth Factor- Hair Serum for the Prevention of Chemotherapy Induced Alopecia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1911187141
Record Dates: First submitted 2020-08-05; First posted 2020-09-18 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Alopecia; Chemotherapy-Induced Change; Hair Loss; Alopecia Drugs
Keywords: Chemotherapy-induced hair loss; Keratinocyte Growth Factor; KGF; Hair loss; Alopecia
MeSH Terms: conditions — Alopecia | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Part 1 - Initial group treatment (Experimental): For part 1 of the study, subjects will be enrolled into a prospective single arm phase where all of them get the study treatment. We plan to enroll up to 25 subjects to have 20 evaluable subjects to this phase.
  Interventions: Drug: Keratinocyte growth factor

INTERVENTIONS:
Drug: Keratinocyte growth factor — At the end of 4 cycles of chemotherapy, primary efficacy end point data will be collected. After 20 evaluable subjects if ≥ 4 responses were noted, part 2 of the study will be activated. The decision rule is based on the lower bound of a one-sided 95% confidence interval; at least 4 out of 20 patients with response results in a lower bound greater than 5% success. The proportion with success and the lower bound of a one-sided exact confidence interval will be computed.

SUMMARY:
Primary aim is to provide a preliminary assessment of the efficacy of the investigational topical formula, KGF-HS, as a prophylactic treatment for chemotherapy induced alopecia.

Hypothesis: KGF-HS will result in less than 50% hair loss by the end of 4 cycles of chemotherapy. The investigators will evaluate hair loss using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 alopecia grading scale.

DETAILED DESCRIPTION:
Primary specific aims

1. To provide a preliminary assessment of the efficacy of the investigational topical formula, KGF-HS, as a prophylactic treatment for chemotherapy induced alopecia.

   Hypothesis: KGF-HS will result in less than 50% hair loss by the end of 4 cycles of chemotherapy. The investigators will evaluate hair loss using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 alopecia grading scale.

   Secondary specific aims
2. To estimate hair preservation as assessed by participant and physician.
3. To estimate participant reported comfort.
4. To evaluate quality of life.
5. To evaluate the incidence of adverse events for topical application.
6. To evaluate if topical hair serum results in faster hair growth after completion of chemotherapy in those who had grade 2 or higher alopecia while on chemotherapy
7. To evaluate responses to chemotherapy at time of surgery (for patients undergoing neoadjuvant chemotherapy (NAC))

Study Design: This study is a 2-part trial. For part 1 of the study, subjects will be enrolled into a prospective single arm phase where all of them get the study treatment. Investigators plan to enroll up to 25 subjects to have 20 evaluable subjects to this phase. At the end of 4 cycles of chemotherapy, primary efficacy end point data will be collected. After 20 evaluable subjects if ≥ 4 responses were noted, part 2 of the study will be activated. The decision rule is based on the lower bound of a one-sided 95% confidence interval; at least 4 out of 20 patients with response results in a lower bound greater than 5% success. The proportion with success and the lower bound of a one-sided exact confidence interval will be computed.

Part 2 of the study is a randomized double blind-placebo controlled trial. Investigators plan to randomize 40 subjects 1:1 to this portion. This sample size was selected to provide 82% statistical power to detect an improvement from a 5% response rate in the control arm to a 35% response rate in the treated arm (assuming a one-sided alpha level of 0.05). Primary efficacy end point will be assessed by clinicians who will be independent and unaware of the study treatment. Participant withdrawals from the study will be deemed treatment failures. Secondary efficacy end points are success in hair preservation assessed by participant's clinician and by the participant, use of wigs and/or head wraps; participant-reported comfort; and quality of life (QOL). Comparison of the proportions between the treated and control arms will be performed using a chi-square test; the confidence interval for the difference between the proportions will be estimated. Comparison of differences in mean quality of life scores will be performed using two sample independent t tests. Adverse events will be reported by grade and tabulated. In phase 1 part of the study, the number of patients undergoing NAC and responses at time of surgery will be noted. No formal statistics will be done. In phase 2 part of the study, proportion of patients undergoing neoadjuvant chemotherapy and their responses at time of surgery will be recorded and comparisons will be done by chi-square test. Investigators do not anticipate the study serum to influence response to chemotherapy as there is no significant systemic absorption however since KGF is a cytoprotective agent, investigators will collect data on response to chemotherapy (for patients undergoing neoadjuvant treatment only).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with early stage breast cancer (stage I-III)
2. Scheduled but not begun, at least 4 cycles of taxane and/or anthracycline-based chemotherapy
3. ≥ 21 years of age
4. Able to give informed consent

Exclusion Criteria:

1. Female pattern hair loss or hair loss disorder
2. Scalp folliculitis
3. Scalp psoriasis
4. Seborrheic dermatitis
5. Inflammatory scalp conditions such as lichen plano-pillaris
6. Subjects wearing wigs or subjects who shave their hair prior to chemotherapy
7. Unable to provide consent or make allotted clinical visits
8. Known allergy to KGF-HS being use in this study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Part 1: Preliminary assessment of the efficacy of the investigational topical formula, KGF-HS measuring hair loss after chemotherapy. | Four months
  Hypothesis: KGF-HS will result in less than 50% hair loss by the end of 4 cycles of chemotherapy. We will evaluate hair loss using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 alopecia grading scale: Grade 1 = Hair loss of <50% of normal; Grade 2 = Hair loss of >50% of normal.
Part 2: Randomized, placebo-controlled assessment of the efficacy of the investigational topical formula, KGF-HS measuring hair loss after chemotherapy. | Four months
  To provide a preliminary assessment of the efficacy of the investigational topical formula, KGF-HS, as a prophylactic treatment for chemotherapy induced alopecia.
  Hypothesis: KGF-HS will result in less than 50% hair loss by the end of 4 cycles of chemotherapy. We will evaluate hair loss using the CTCAE (Common Terminology Criteria for Adverse Events) v4.0 alopecia grading scale: Grade 1 = Hair loss of <50% of normal; Grade 2 = Hair loss of >50% of normal.

SECONDARY OUTCOMES:
Hair preservation as assessed by participant. | Four months
  To estimate hair preservation using the Alopecial Pictoral Tool in Appendix A of protocol. Grades 0-2 per CTCAE v4.0.
Hair preservation as assessed by physician. | Four months
  To estimate hair preservation using the Alopecial Pictoral Tool in Appendix A of protocol. Grades 0-2 per CTCAE v4.0.
Estimate participant reported comfort. | Four months
  To estimate participant reported comfort using the Comfort Scale from Massey study 2004 as found in Appendix B of protocol. Ratings on a scale from Very Comfortable through Very Uncomfortable.
Evaluate quality of life using EORTC QLQ-C30 | Four months
  The emotional functional scale score is calculated from EORTC QLQ Q30 items 21-24 and the social functioning scale is calculated from EORTC QLQ-C30 items 26 and 27 using the EORTC QLQ-C30 scoring formula, which linearly transformed the average raw scored to a range from 0 to 100 (a higher score represented a higher level of functioning).
  The BIS summary score will be the sum of the first 9 (of 10) items in the BIS.
Evaluate quality of life using HADS. | Four months
  The HADS (Hospital Anxiety and Depression Scale) will be used to assess anxiety and depression. It includes 7 questions to assess anxiety and 7 to assess depression. The summary scores (sum of the 7 question items) for anxiety and depression range from 0 to 21: scores of 0 to 7 are considered normal, 8 to 10 are considered borderline abnormal (borderline case), and 11 to 21 are considered abnormal (case). Missing items will be replaced by the average of non-missing items if only 1 item from the anxiety or depression scale was missing.
Evaluate quality of life using BIS. | Four months
  The BIS (Body Image Scale) summary score will be the sum of the first 9 (of 10) items in the BIS. The last item in the BIS for scar is not applicable to the study participants, so it will not be included. The summary score ranges from 0 to 27; a score of 0 indicates no symptoms or distress, and a higher score indicated increasing symptoms or distress. Missing items will be replaced by the average of non-missing items if only 1 or 2 items from the 9 items in the BIS are missing.
Evaluate the incidence of adverse events for topical application. | Four months
  To evaluate the incidence of adverse events for topical application.
Evaluate hair regrowth. | Four months
  To evaluate if topical hair serum results in faster hair growth after completion of chemotherapy in those who had grade 2 or higher alopecia while on chemotherapy compared to control group.Using the Alopecial Pictoral Tool in Appendix A of protocol. Grades 0-2 per CTCAE v4.0.
Evaluate responses to chemotherapy at time of surgery. | Four months
  To evaluate responses to chemotherapy at time of surgery (for patients undergoing neoadjuvant chemotherapy (NAC)) as assessed by physician through pathology measuring tumor size at site.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States